CLINICAL TRIAL: NCT02466204
Title: An Efficacy and Safety Study of Corifollitropin Alfa Versus Daily Follitropin Beta for Controlled Ovarian Stimulation in Women 35-42 Years Old With a Body Weight ≥ 50 kg Undergoing IVF Treatment.
Brief Title: Efficacy of Corifollitropin Alfa Versus Follitropin Beta in Aged IVF (In-vitro Fertilization) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_ 01_2015
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- corifollitropin alfa (long action FSH) (Active Comparator): corifollitropin alfa 150 mcg subcutaneous injection. Seven days after, combines with recombinant FSH 300 IU daily subcutaneous injection
  Interventions: Drug: corifollitropin alfa
- Follitropin Beta (recombinant FSH) (Active Comparator): 300 IU of recombinant FSH, daily subcutaneous injection
  Interventions: Drug: Follitropin Beta

INTERVENTIONS:
Drug: corifollitropin alfa — Drug is injected subcutaneously. Seven days after, 300 IU FSH daily injected subcutaneously, until at least two leading ovarian follicles reach 17mm in diameter.
  Other Names: Elonva
  Arms: corifollitropin alfa (long action FSH)
Drug: Follitropin Beta — Drug is injected subcutaneously, daily, until at least two leading ovarian follicles reach 17mm in diameter.
  Other Names: Puregon
  Arms: Follitropin Beta (recombinant FSH)

SUMMARY:
A prospective, randomized, controlled study to explore the efficacy and safety of using either corifollitropin alfa 150 mcg or daily recombinant follicle stimulation hormone (FSH) 300 international unit (IU) for the stimulation treatment of subjects undergoing controlled ovarian stimulation prior to IVF.

The study is designed as a non-inferiority trial. The sample size for this trial of 400 subjects, in both groups, being treated for one IVF cycle is based upon the primary endpoint of the number of oocytes retrieved.

DETAILED DESCRIPTION:
Stimulation regimen and assisted reproductive technology procedures

Corifollitropin Alfa Group: On day 2 or day 3 of the menstrual cycle, a single subcutaneous injection of corifollitropin alfa 150 mg/ 0.5 mL is administered (stimulation day 1).

FSH Group: Daily subcutaneous injections with recombinant FSH (Follitropin Beta) 300 international units (IU) is started on On day 2 or day 3 of the menstrual cycle (stimulation day 1) and continue up to and including stimulation day 7.

From stimulation day 8 onwards, subjects from both treatment groups will continue with a daily subcutaneous dose of FSH up to the day before human chorionic gonadotropin (hCG) administration or gonadotropin releasing hormone agonist administration day. The maximum FSH dose to continue treatment after the first 7 days is 300 IU, but the dose could be reduced when desired.

To prevent premature luteinizing hormone (LH) surges the gonadotropin releasing hormone (GnRH) antagonist (ganirelix acetate subcutaneous injection, 0.25 mg/ 0.5 mL) is administered, starting on stimulation day 5.

As soon as at least three follicles of 17 mm are observed by ultrasound, hCG or a GnRH agonist will be used for final oocyte maturation at the same day. hCG is used if 3-18 follicles and 0.2 mg triptorelin is administered if ≥ 19 follicles >11 mm are observed. About 34-36 hours thereafter, oocyte retrieval followed by IVF or intra-cytoplasmic sperm injection (ICSI) is performed. Three days after oocyte pick-up, 2 to 3 fresh embryos will be transferred. If patients have high progesterone level on day of trigger (progesterone level > 1,5 ng/ml), risk of OHSS and unfavorable endometrium, fresh transfers will be cancelled and freeze all will be recommended.

Patients using hCG for final oocyte maturation will receive luteal phase support with progestogen gel (90 mg once daily) intra-vaginally and estradiol (4 mg/day orally, twice daily) initiated on the day of oocyte retrieval or the day thereafter. Patients, using GnRH agonist for triggering, will have fresh transfer with intense luteal phase support of estradiol and progesterone (receive intense luteal phase support with estradiol and progesterone as the same dose mentioned above and progesterone 50 mg intramuscular injection per day).

Assessments

Patients will return to the clinic for pregnancy test 2 weeks after embryo transfers.

Local tolerance parameters (pain, itching, swelling and redness) are assessed by the clinical staff 30 min after injection for both corifollitropin alfa and FSH injection sites.

Clinical Outcome The primary objective is to show that the corifollitropin alfa regimen, in terms of the number of oocytes retrieved, is equivalent to the reference treatment (predefined equivalence range: -3 to +5 oocytes).

Other clinical parameters will also be evaluated: dose of FSH required, duration of stimulation, number and size of follicles (≥11mm and ≥14 mm), serum hormone levels, fertilization rate, number and quality of embryos obtained, implantation rate, miscarriage rate, and pregnancy rates.

At least 14 days after embryo transfer, a blood pregnancy test is performed. If the pregnancy test is positive, vaginal and/or abdominal ultrasonographic investigation is performed between 35 and 42 days ( 5 to 6 weeks) after embryo transfer to confirm a clinical pregnancy and at least 70 days (≥ 10 weeks) after embryo transfer to confirm an ongoing pregnancy.

Patients will be followed to one year after randomization.

All efficacy analyses will be based on the intent-to-treat (ITT) population, which included all randomized patients who will receive corifollitropin alfa or at least one dose of FSH

Safety endpoints

Occurrence of adverse events, including moderate and severe ovarian hyperstimulation syndrome (OHSS), outcome of local tolerance at injection site assessments will be evaluated as safety endpoints.

The percentage of patients with moderate or severe OHSS and local tolerance is compared between the treatment groups using Fisher's exact test.

Safety analyses will be performed on the all-subjects-treated group, which comprised all the patients who will receive either corifollitropin alfa or FSH.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be willing and able to provide written informed consent for the study.
* Each subject must be female with years of age ≥35 to ≤42 at the time of recruitment..
* Each subject must have an indication for controlled ovarian stimulation and IVF
* Each subject must have a body weight ≥ 50.0 kg, with a body mass index (BMI) ≥18.0 to ≤32.0 kg/m2.
* Each subject must have a regular spontaneous menstrual cycle with an intra-individual variation not outside the 24 to 35 days range.
* For each subject, ejaculatory sperm must be available (use of donated and/or cryopreserved sperm is allowed; sperm obtained via surgical sperm retrieval is not allowed).
* Each subject must have results of clinical laboratory test (complete blood count, blood chemistries, and urinalysis) within normal limits or clinically acceptable to the investigator, as measured by the local laboratory at screening. A normal cervical smear result, obtained within 12 months, otherwise it must be obtained during screening.
* Each subject must have results of a physical examination, including blood pressure, within normal limits or clinically acceptable limits to the investigator.
* Each subject must have normal ovarian reserve, based on anti-Mullerian hormon (AMH) of 1.38 - 3.25ng/ml or an antral follicle count (AFC) of 7-20, taken within 2 months prior to corifollitropin alfa start.
* Each subject must be able to adhere to dose and visit schedules and willing to disclose any medical events to the investigator.

Exclusion Criteria:

* The subject has a recent (ie, within 3 years) history of/ or any current endocrine abnormality (irrespective whether the patient is stabilized on treatment).
* The subject has a history of ovarian hyper-response (ie, previous IVF cycle with more than 30 follicles ≥11 mm on ultrasound) or ovarian hyperstimulation syndrome (OHSS).
* The subject has a history of/or current polycystic ovary syndrome (PCOS)
* The subject has more 20 basal antral follicles <11 mm (both ovaries combined) as measured on ultrasound in the early follicle phase (menstrual cycle day 2-5).
* The subject has less than 2 ovaries in any other ovarian abnormality (including endometrioma > 10 mm; visible on ultrasound).
* The subject has unilateral or bilateral hydrosalpinx (visible on ultrasound, less clipped).
* The subject has any intra-uterine fibroids >5 cm or any clinically relevant pathology, which could impair embryo implantation or pregnancy continuation.
* The subject has more than three unsuccessful treatment cycles for IVF/ICSI.
* The subject has a history of non- or low avarian response to FSH / Human Menopausal Gonadotropin (hMG) treatment (ie, previous COS cycle cancelled due to insufficient ovarian response or ≤3 oocytes obtained).
* The subject has a history of current miscarriage (3 or more, even when explained).
* The subject has FSH > 15.0 IU/L or LH > 12 .0 IU/L as measured by the local laboratory (sample taken during the early follicle phase: menstrual cycle day 2 to 5).
* The subject has tested positive for human immunodeficiency virus (HIV) or Hepatitis B (results obtained within one year) .
* The subject has contra-indications for the use of gonadotropins (eg, tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, or ovarian cysts) or GnRH antagonist (eg, hypersensitivity, pregnancy/lactation).
* The subject has a concomitant use of either LH or hMG/urinary FSH preparations in study cycle.
* The subject has a recent history of/or current epilepsy, thrombophilia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary or auto-immune disease requiring regular treatment.
* The subject or the sperm donor has known gene defects, genetic abnormalities, or abnormal karyotyping, relevant for the current indications or for the health of the offspring.
* The subject smokes or has recently stopped smoking (ie, within the last 3 months prior to signing ICF).
* The subject has a history or presence of alcohol or drug abuse within 12 months prior to signing informed consent.
* The subject has an allergy/ sensitivity to investigational drugs or their excipients.
* The subject has used any experimental drugs within 3 months prior to signing informed consent.
* The subject is participating in any other clinical study (excluding surveys).

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
number of oocytes | 10 minutes after oocyte retrieval completed
  in 10 minutes after oocyte retrieval, total number of oocytes retrieved is counted and recorded

SECONDARY OUTCOMES:
Rate of moderate and severe ovarian hyperstimulation syndrome | 8 days after oocyte retrieval
  symptoms of ovarian hyperstimulation syndrome are followed and recorded until 8 days after oocyte retrieval.
Live birth | at the time of delivery
  delivery of live birth
number of MII oocytes | 2 hours after oocyte retrieval completed
  Number of mature oocytes collected
number of 2PN | 18 hours after sperm injection
  number of two pronuclear (2PN) fertilized oocytes
number of mature follicles >11 mm | on the day of hCG administration
  number of mature follicles >11 mm in diameter
estradiol level | on the day of hCG administration
  serum level of estradiol
FSH dose | calculated on the day of hCG administration
  total dose of FSH
implantation rate | 5 to 6 weeks after embryo transfer
  number of sacs with heart beat per total number of embryos transferred
Clinical pregnancy | at 5 to 6 six weeks after embryo transfer
  gestational sac on ultrasound
Ectopic pregnancy | 7 to 8 weeks after embryo transfer
  The presence of a gestational sac outside the uterine cavity shown on sonography or laparoscopy
Miscarriage | 7 to 12 weeks of gestation
  Loss of clinical pregnancy
Multiple pregnancy | at 7 weeks of gestation
  more than one gestational sacs or heart beats on ultrasound
Ongoing pregnancy | at 10 weeks after embryo transfer
  At least one gestational sac on ultrasound
Cumulative ongoing pregnancy | at 12 months after randomization
  Cumulative ongoing pregnancy at 12 months after randomization
Pregnancy-induced hypertension | measured at or after 20 weeks gestation
  systolic blood pressure ≥140 mmHg or diastolic pressure ≥90 mmHg on two occasions, two hours apart, or severely elevated single blood pressure measurement requiring antihypertensive medication
Pre-eclampsia | measured at or after 20 weeks gestation
  hypertension plus proteinuria or other organ involvement, neurologic or hematologic complications, uteroplacental dysfunction, or fetal growth restriction
HELLP syndrome | measured at or after 20 weeks gestation
  Elevated liver enzyme levels (aspartate aminotransferase ≥100 U/L), thrombocytopenia (platelet count <100,000/mm3), elevated serum creatinine level (≥1.5 mg/dL [132.6 μmol/L]) and/or hemolysis (hemoglobin <10 g/dL)
Gestational diabetes mellitus | measured at or after 20 weeks gestation
  Diagnosed using a 75g oral glucose tolerance test; fasting: 92 mg/dL [5.1 mmol/L]; 2-hour: 153 mg/dL [8.5 mmol/L]
Prematurity | at 24 weeks gestation, at 32 weeks gestation, at 34 weeks gestation, and at 37 weeks' gestation
  preterm birth if any
Cumulative live birth | at 12 months after randomization
  cumulative live birth delivery at 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - My Duc Hospital, Ho Chi Minh City
  - Research Center for Genetics and Reproductive Health, Ho Chi Minh City

REFERENCES:
- [Derived] Vuong NL, Pham DT, Phung HT, Giang HN, Huynh GB, Nguyen TTL, Ho MT. Corifollitropin alfa vs recombinant FSH for controlled ovarian stimulation in women aged 35-42 years with a body weight >/=50 kg: a randomized controlled trial. Hum Reprod Open. 2017 Nov 28;2017(3):hox023. doi: 10.1093/hropen/hox023. eCollection 2017. PMID 30895237